CLINICAL TRIAL: NCT05542940
Title: P53 Immunohistochemistry Abnormal Staining in Endometrial Cancer and Its Relation With Disease Stages, Pathological Types and Grading
Brief Title: P53 Immunohistochemistry Abnormal Staining in Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Hossam Hassan Aly Hassan El Sokkary (Other)
Responsible Party: Sponsor-Investigator, Hossam Hassan Aly Hassan El Sokkary, Associate professor, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: SOKKARY9
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: p 53 immunohistochemistry positive staining and relation to stages ,pathological types and grading — p 53 immunohistochemistry positive staining and relation to stages ,pathological types and grading

SUMMARY:
Objective: Calculate the incidence of P53 immunohistochemistry abnormal staining in endometrial cancer and to identify its relation with disease stages, pathological types and grading.

Patients and methods:

100 cases of endometrial cancer will be included in the study, recruited from Alexandria university hospital gyne-oncology unit. Surgical staging, histopathological examination and immunohistochemistry of p53 were done to all cases to calculate the incidence of P53 immunohistochemistry abnormal staining in endometrial cancer and to identify its relation with disease stages, pathological types, grading.

Keywords: P53 immunohistochemistry, endometrial cancer, clinicopathological relation.

ELIGIBILITY:
Inclusion Criteria:

* endometrial cancer patients

Exclusion Criteria:

* patients unfit for surgery

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: randomized
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
p53 immunohistochemistry | 1 month
  Incidence of abnormal staining of p53 in endometrial cancer
Relation of p53 abnormal staining with disease stages | 1month
  Relation of p53 abnormal staining with disease stages
Relation of p53 abnormal staining with disease pathological types | 1 month
  Relation of p53 abnormal staining with disease pathological types
Relation of p53 abnormal staining with disease pathological grades | 1 month
  Relation of p53 abnormal staining with disease pathological grades

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam Hassan El Sokkary, Alexandria, Egypt